CLINICAL TRIAL: NCT03454711
Title: Functional Magnetic Resonance Imaging (fMRI) Exploration of Neurocognitive Processes Involved in Food Addiction (FA) in Obese Patients: Towards New Phenotypic Markers for an Optimized Care Pathway
Acronym: AddictO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Institut NuMeCan, INRAE 1341 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC17_8949_AddictO; 2017-A01269-44 (Other: N°ID-RCB)
Record Dates: First submitted 2018-02-20; First posted 2018-03-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Obesity; Food addictions; Functional magnetic resonance imaging (fMRI); Metabolomics
MeSH Terms: conditions — Obesity; Food Addiction | interventions — Magnetic Resonance Imaging; Calorimetry, Indirect; Glucose; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with food addcitions (Experimental): Patients (20) will be selected from the Yale Food Addiction Scale (YFAS): a validated screening of FA questionnaire.
  Three clinical visits will be realized in less than two months
  Interventions: Device: fMRI; Device: Indirect calorimetry; Device: Bioimpedance; Biological: Lipid profile, glucose, HBA1c, metabolomic analysis; Behavioral: YFAS questionnaire, Binge Eating Scale, Hospital Anxiety and Depression (HAD) scale, hedonic evaluation test (liking)
- Patients without food addictions (Experimental): Patients (20) will be selected from the Yale Food Addiction Scale (YFAS): a validated screening of FA questionnaire.
  Three clinical visits will be realized in less than two months
  Interventions: Device: fMRI; Device: Indirect calorimetry; Device: Bioimpedance; Biological: Lipid profile, glucose, HBA1c, metabolomic analysis; Behavioral: YFAS questionnaire, Binge Eating Scale, Hospital Anxiety and Depression (HAD) scale, hedonic evaluation test (liking)

INTERVENTIONS:
Device: fMRI — Brain MRI
Device: Indirect calorimetry — Resting energy expenditure
Device: Bioimpedance — Measurement of body composition
Biological: Lipid profile, glucose, HBA1c, metabolomic analysis — Blood sample
Behavioral: YFAS questionnaire, Binge Eating Scale, Hospital Anxiety and Depression (HAD) scale, hedonic evaluation test (liking) — Questionnaires to characterize eating habits and depression

SUMMARY:
Identification of the cerebral fMRI phenotype of obese patients with FA in cognitive task context based on food choice making

DETAILED DESCRIPTION:
Obesity is a worldwide epidemic associated with many complications. The treatment of obesity is a failure if it does not take into account eating disorders. Among them, food addictions seem to be frequent among obese patients. Clinical diagnosis and therapeutic approaches depend on presence of these FA. Moreover, eating disorders are associated with visible brain abnormalities in fMRI but the cerebral fMRI phenotype of FA is not known.

ELIGIBILITY:
Inclusion Criteria:

* female
* right-handed
* grade 1 and 2 obesity
* aged between 20 and 50
* no other addictions including smoking
* no contraindications to fMRI
* affiliated to French Social Security
* having given a written informed consent

Exclusion Criteria:

* abdominal circumference + upper limbs along the body > 200cm
* addiction to alcohol or other psychoactive substances
* daily smoker
* sleep Apnea Syndrome paired
* psychotic psychiatric disorders
* history of bariatric surgery
* medical care in the nutrition unit
* inability to comprehend or complete questionnaires
* pregnant or breastfeeding woman
* persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Significant change in brain activity of the prefrontal cortex (area involved in the inhibitory control of food intake) measured by modification of BOLD (Blood-Oxygen-Level-Dependent) signal in fMRI during a cognitive task based on food choice making | Month 2

CONTACTS AND LOCATIONS:
Overall Officials: David Val-Laillet, MSc, PhD, HDR, Study Director — Institut NuMeCan, INRA 1341, INSERM 1241, Université de Rennes 1
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No